CLINICAL TRIAL: NCT02522793
Title: Non-Invasive Optical Spectroscopy for Identification of Cutaneous Cancer
Brief Title: Optical Spectroscopy for Cutaneous Cancer
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00058440
Record Dates: First submitted 2015-08-12; First posted 2015-08-13 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Suspicious Skin Lesion(s) Requiring a Biopsy
Keywords: skin lesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention; this is an observational study

SUMMARY:
1. Purpose and objective: Determine spectroscopic differences between tumor, dysplasia, and normal cutaneous tissue as assessed by histopathologic diagnosis. If successful, the optical measurements could be used to survey for and delineate the extent of malignancies in a noninvasive manner.
2. Study activities and population group: Competent adults with a clinically suspicious skin lesion who are undergoing a biopsy as part of their routine care. For those who agree to participate, the sterilized portable optical spectroscopic probe will be used to measure diffuse reflectance on the lesion of clinical interest.
3. Data analysis and risk/safety issues: The optical spectrometer does not breach any skin defense barrier. As this study involves noninvasive optical measurements of tissues, no significant safety concerns are anticipated. Qualitative analysis will be performed to describe whether there is correlation between spectroscopy measurements and pathologic diagnosis. A variety of correlative statistics will be explored to determine if there are relationships found that can justify a larger study

DETAILED DESCRIPTION:
This is a pilot study to determine the optical spectroscopy characteristics of tumor in patients with cutaneous malignancies. These spectroscopy measurements will be compared with pathological diagnosis of tissue biopsies from the same site. If successful, the optical measurements could be used to survey for and delineate the extent of malignancies in a noninvasive manner. This would be especially helpful for clinic visits where suspicious lesions are seen and would otherwise require biopsy for diagnosis. Immediate benefits would include patients with numerous suspicious skin lesions who would require multiple biopsies.

Further spectroscopy measurements of the tumor site and adjacent normal tissue during therapy (chemoradiotherapy or radiotherapy) may provide useful information pertinent to tumor physiology and therapeutic effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one clinically suspicious skin lesion warranting a biopsy as part of routine care, in the outpatient clinic setting.
* Patients with previous histologically confirmed malignancy such as basal cell carcinoma or squamous cell carcinoma are eligible; however this is not required for enrollment.
* The suspicious skin lesion(s) is accessible to optical probe measurements. If patient has previous histologically confirmed malignancy of the skin, then the primary tumor site must be accessible to optical probe measurements
* Patient is able to provide written informed consent
* Patient is >18 years of age

Exclusion Criteria:

* < 18 years of age
* Unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to the Duke or VA Dermatology or Otolaryngology clinics with a suspicious skin lesion that is in need of a biopsy.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-02-03 (Actual); Study Completion 2017-02-03 (Actual)

PRIMARY OUTCOMES:
spectroscopic differences between tumor, dysplasia, and normal cutaneous tissue. | 1 day visit
  Determine spectroscopic differences between tumor, dysplasia, and normal cutaneous tissue as assessed by histopathologic diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Woodard, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States